CLINICAL TRIAL: NCT05805306
Title: Promoting HIV PrEP Among MSM: a Randomized Control Trial - Aim 3
Brief Title: Entre Herman@s: Promoting Health Among Latino MSM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: St. Johns Community Health (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Homero del Pino, Associate Professor, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1995640-1; U54MD007598 (NIH)
Record Dates: First submitted 2023-03-01; First posted 2023-04-10 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections
Keywords: Men Who Have Sex with Men; Latino men; HIV PrEP; Siblings
MeSH Terms: conditions — HIV Infections; Homosexuality | interventions — Vaccines; Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP Promotion (Experimental)
  Interventions: Behavioral: Entre Herman@s
- Vaccine Promotion (Placebo Comparator)
  Interventions: Behavioral: Vaccines for Health

INTERVENTIONS:
Behavioral: Entre Herman@s — The intervention unfolds as follows: (Week 1) the research team, Latino MSM, & sibling will all engage in a PrEP Conversation followed by an individual Sibling Training for siblings to learn communication strategies for promoting health behaviors; (Week 2) we will send siblings reminders and a link to motivational interviewing techniques; (Week 3) we will conduct brief Follow-ups with siblings to determine if their brother changed his behavior; (Week 4) we will send a reminder to Latino MSM that they will have a follow-up the following week; (Week 5) we will conduct 30-day Follow-up with Latino MSM to determine if there was uptake of the new behavior change; (Week 7) same as week 5 above; (Week 10) send siblings information on motivational interviewing; (Week 12) final follow-up for both Latino MSM and siblings.
  Arms: PrEP Promotion
Behavioral: Vaccines for Health — The intervention unfolds as follows: (Week 1) the research team, Latino MSM, & sibling will all engage in a Health Conversation about vaccines for COVID, Hep A/B, or MPOX, followed by an individual Sibling Training for siblings to learn communication strategies for promoting health behaviors; (Week 2) we will send siblings reminders and a link to motivational interviewing techniques; (Week 3) we will conduct brief Follow-ups with siblings to determine if their brother changed his behavior; (Week 4) we will send a reminder to Latino MSM that they will have a follow-up the following week; (Week 5) we will conduct 30-day Follow-up with Latino MSM to determine if there was uptake of the new behavior change; (Week 7) same as week 5 above; (Week 10) send siblings information on motivational interviewing; (Week 12) final follow-up for both Latino MSM and siblings.
  Arms: Vaccine Promotion

SUMMARY:
This is a randomized controlled trial with an attention placebo control group. The goal of this study is to decrease HIV incidence in Latino men who have sex with men by engaging their siblings in PrEP-use promotion. In the intervention arm, siblings will be trained to engage their gay brother in PrEP conversations. In the control arm, siblings will be trained to engage their gay brother in conversations about vaccines to prevent COVID, Hepatitis A/B, or MPOX.

ELIGIBILITY:
Inclusion Criteria: Latino Men Who Have Sex with Men

1. self-identify as Latino
2. identify as male
3. be <40 years old
4. report HIV-negative status
5. be willing to talk about MSM healthcare issues with a sibling
6. either (a) have never used PrEP or (b) stopped using PrEP at least 90 days ago
7. missing most recent COVID vaccine
8. missing Hepatitis (A or B) vaccines
9. missing Mpox vaccine
10. meet CDC's PrEP eligibility criteria (be HIV-negative; any male sex partner in the past six months; not in a monogamous partnership with a recently tested, HIV-negative man; and at least one of the following: any anal sex without condoms in past 6 months, any sexually-transmitted infection (STI) diagnosed or reported in past 6 months, or is in an ongoing sexual relationship with an HIV-positive male partner).

Exclusion Criteria: Latino Men Who Have Sex with Men

1. are unable to provide consent or
2. they do not meet any of the criteria above

Inclusion Criteria: Siblings

1. at least 18 years old
2. report a close relationship his/her LMSM brother <40 years old
3. be willing to talk about MSM healthcare issues with his/her LMSM brother

Exclusion Criteria: Siblings

1. are unable to provide consent or
2. they do not meet any of the criteria above

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2023-04-29 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants that start using PrEP | 90 days
  This measures how many participants in the experiment group started taking PrEP (baseline = 0 participants).
  Tool: Pictures. Participants will submit a picture of their pill bottle to report PrEP use.
Number of participants that get vaccinated | 90 days
  This measures whether participants in the control group decided to get vaccinated for COVID, Hep A/B, or MPOX.
  Tool: Pictures. Participants will submit a picture of their proof-of-vaccination card to report vaccination status.

SECONDARY OUTCOMES:
Number of participants who increase their willingness to use PrEP | 90 days
  This measures whether participants progress along the stages of change (e.g., pre-contemplation, contemplation, action) in their willingness to try PrEP if it were available to them.
  Tool: Stages of Change questionnaire administered at baseline and 90 days.
Number of participants who increase their willingness to get vaccinated | 90 days
  This measures whether participants progress along the stages of change (e.g., pre-contemplation, contemplation, action) in their willingness to get vaccinated against COVID, Hep A/B, or MPOX if it were available to them.
  Tool: Stages of Change questionnaire administered at baseline and 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Homero del Pino, PhD, MS, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles R. Drew University of Medicine and Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No